CLINICAL TRIAL: NCT02153060
Title: A Multi-center, Randomized, Open-label Study to Evaluate the Efficacy and Safety of Different Doses of Dexamethasone for Management of Immune Thrombocytopenia (ITP)
Brief Title: An Investigation of Dexamethasone With Different Doses in the Management of Immune Thrombocytopenia (ITP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); Shandong Provincial Hospital (Other Government); The First Affiliated Hospital of Dalian Medical University (Other); Peking Union Medical College Hospital (Other); Shandong University of Traditional Chinese Medicine (Other); Anhui Provincial Hospital (Other Government); Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Dexamethasone
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2014-05

CONDITIONS: Immune Thrombocytopenia
Keywords: immune thrombocytopenia; dexamethasone; efficacy; safety
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20mg dexamethasone group (Experimental): Dexamethasone 20 mg per day, 4 consecutive days
  Interventions: Drug: Dexamethasone
- 40mg dexamethasone group (Experimental): Dexamethasone 40 mg per day, 4 consecutive days
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone was given at a dose of 40 mg,daily for 4 consecutive days
  Arms: 40mg dexamethasone group
Drug: Dexamethasone — Dexamethasone was given at a dose of 20 mg,daily for 4 consecutive days
  Arms: 20mg dexamethasone group

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University and other 7 well-known hospitals in China. In order to report the efficacy and safety of different dose dexamethasone in treating the immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicentre, randomised controlled trial of 60 adults with ITP from 7 medical centers in China. Part of the participants are randomly selected to receive dexamethasone (given at a dose of 40mg per day for 4 consecutive days) ,the others are selected to receive dexamethasone(given at a dose of 20 mg daily for 4 days).

Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study. In order to report the efficacy and safety of different dose dexamethasone for the treatment of adults with immune thrombocytopenia (ITP).

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia
2. Untreated hospitalized patients, may be male or female, between the ages of 18 ~ 75 years
3. To show a platelet count <30 * 10^9/L, and with bleeding manifestations
4. Willing and able to sign written informed consent

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit
2. Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit
3. Received high-dose steroids or IVIG in the 3 weeks prior to the start of the study
4. Current HIV infection or hepatitis B virus or hepatitis C virus infections
5. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
6. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period
7. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test
8. Patients who are deemed unsuitable for the study by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Proposed criteria for assessing early response to ITP treatments | 3 months
  1. Complete response (CR)： A platelet count ≥ 100 * 10^9/L measured on two occasions > 7 days apart and the absence of bleeding.
  2. Response (R)： A platelet count ≥ 30 * 10^9/L and a greater than two fold increase in platelet count from baseline measured on two occasions > 7 days apart and the absence of bleeding.
  3. No response (NR)： A platelet count < 30 * 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.

SECONDARY OUTCOMES:
Safety | 1 years
  The type and frequency of therapy associated adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, DR., Principal Investigator — Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Background] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889
- [Background] Cheng Y, Wong RS, Soo YO, Chui CH, Lau FY, Chan NP, Wong WS, Cheng G. Initial treatment of immune thrombocytopenic purpura with high-dose dexamethasone. N Engl J Med. 2003 Aug 28;349(9):831-6. doi: 10.1056/NEJMoa030254. PMID 12944568